CLINICAL TRIAL: NCT04161092
Title: A Randomized Controlled, Open-label, Multicentre Study Evaluating if Liver Transplantation With Liver Grafts From Extended Criteria Donors Not Utilised for Approved Indications Increases Overall Survival in Patients With Non-resectable Isolated Liver Metastases From Colorectal Metastases, in Comparison With Best Alternative Care
Brief Title: The Swedish Study of Liver Transplantation for Non-resectable Colorectal Cancer Metastases
Acronym: SOULMATE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOULMATE
Record Dates: First submitted 2019-10-31; First posted 2019-11-13 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Cancer; Liver Metastases; Colorectal Liver Metastases
Keywords: colorectal cancer; liver metastases; liver transplant; non-resectable colorectal cancer metastases
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liver transplantation + best alternative care (Other): Patients subjected to Ltx will during the waiting time receive individualized chemotherapy, with the aim to avoid side effect that make them not transplantable.
  If possible, patients randomized to Ltx should be treated within 12 weeks after randomization.
  If the patients progress systemically they will be treated with best alternative care.
  If they progress only within the liver they continue to be transplantable until they are deemed technically not transplantable by the transplant surgeon.
  Interventions: Procedure: Liver transplantation Ltx
- Best alternative care (Other): The treating physician will together with the patient decide the treatment.
  Interventions: Other: Best alternative care

INTERVENTIONS:
Procedure: Liver transplantation Ltx — Patients will be treated with Ltx at Sahlgrenska University Hospital, Göteborg, or Karolinska University Hospital, Huddinge.
  Arms: Liver transplantation + best alternative care
Other: Best alternative care — All available treatments as well as other experimental treatments are tolerated, however no cross-over to other arm will be allowed.
  Arms: Best alternative care

SUMMARY:
To evaluate if the addition of liver transplantation primarily utilizing liver grafts from extended criteria donors not utilized for approved indications to conventional treatment of non-resectable/ non-abatable colorectal liver metastases (CLM) increases overall survival compared to best alternative care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-resectable, non-ablatable liver metastases from colorectal adenocarcinoma.
* Male or female 18 years or above.
* Primary tumour removed with an R0 resection, and histologically verified adenocarcinoma from colon or rectum
* Liver metastases measurable by MRI or CT according to RECIST version 1.1 Imaging within 4 weeks prior to inclusion.
* No signs of extrahepatic metastatic disease or local recurrence according to MRI and CT of thorax/abdomen and whole body Positron-emission tomography (PET)/ computed tomography (CT) scan.
* A colonoscopy performed within the last 12 months in order to exclude multifocal colorectal cancer (CRC) tumours.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Satisfactory blood tests: Hb ≥ 90 g/L (transfusions are permitted to achieve baseline hemoglobin level), White blood cell Count (WBC) >3,0x109/L, Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L, platelet Count (PLT) >75, Bilirubin<2 x upper normal level, Aspartate aminotransferase (ASAT), Alanine aminotransferase (ALAT)<5 x upper normal level, Calculated Creatinine clearance ≥ 50 mL/min(MDRD).
* Received at least 2 months of chemotherapy with no signs of progressive disease according to RECIST-criteria at the last evaluation before randomization.
* One year or more from the initial CRC diagnosis to the date of inclusion in the study
* Patient accepted for transplantation by a national study board
* Signed and dated written informed consent before the start of specific protocol procedures.

Exclusion Criteria:

* Evidence of extrahepatic disease by PET-CT or CT-thorax/abdomen.
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within seven days prior to the start of study.
* Weight loss >10% the last 6 months
* Other malignancies within the last 5 years, except CRC and low risk tumours such as basaliomas.

  * Liver metastases larger than 10 cm.
* Pathological lymphatic nodes in the abdomen. If a patient has pathological lymphatic nodules in the hepatoduodenal ligament, a staging operation with histo-pathological examination from the nodules with no signs of tumour cell involvement has to be performed before inclusion.
* BRAF (a gene that encodes a protein called b-raf) mutation in primary tumour
* microsatellite instability (MSI-H) in primary tumour
* Previous organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Five-year overall survival | randomization to follow up at 5 years
  Percentage of subject who reach the endpoint of overall survival

SECONDARY OUTCOMES:
Two-year overall survival | randomization to follow up at 2 years
  Percentage of subject who reach the endpoint of overall survival
Median overall survival | : Date of randomization until the date of death from any cause, assessed up to 5 years
  Defined as time to death
Progression-free survival | Date of randomization until the date of documented progression of existing lesions or appearance of new lesions, assessed up to 5 years
  Defined as time from randomization to progress of existing lesions, or appearance of new lesions, within the liver according to RECIST criteria (version 1.1) using CT or MRI and analysed using Kaplan-Meier and the log-rank test.
Hepatic progression-free survival | Date of randomization until the date of documented progression of existing lesions or appearance of new lesions in the liver, assessed up to 5 years
  Defined as time from randomization to progress of existing lesions in the liver , or appearance of new lesions in the liver, according to RECIST criteria (version 1.1) using CT or MRI and analysed using Kaplan-Meier and the log-rank test.
Extrahepatic recurrence-free survival | Date of randomization until the date of documented appearance of new extra-hepatic lesions, assessed up to 5 years
  Defined as time from randomization to appearance of new extra-hepatic lesions, using CT or MRI and analysed using Kaplan-Meier and the log-rank test.
Changes in quality of Life assessed with Euroqol Group Questionaire 5D-3L (EQ-5D-3L) | baseline, 3, 6, 12, 18, 24, 36 and 60 months
  Assessed with EQ-5D-3L
Health economic evaluation | baseline, 3, 6, 12, 18, 24, 36 and 60 months
  Estimation of Quality Adjusted Life Year (QALY) assessed with EQ-5D-3L

CONTACTS AND LOCATIONS:
Overall Officials: Per G Lindner, MD, PhD, Principal Investigator — Transplant Institute, Sahlgrenska University Hospital; Carl Jorns, MD, PhD, Study Director — Transplantation Unit, Karolinska University Hospital
Locations (2):
- Sweden (2):
  - Transplant Institute, Sahlgrenska University Hospital, Gothenburg
  - Transplantation Unit, Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdalla EK, Vauthey JN, Ellis LM, Ellis V, Pollock R, Broglio KR, Hess K, Curley SA. Recurrence and outcomes following hepatic resection, radiofrequency ablation, and combined resection/ablation for colorectal liver metastases. Ann Surg. 2004 Jun;239(6):818-25; discussion 825-7. doi: 10.1097/01.sla.0000128305.90650.71. PMID 15166961
- [Background] Hagness M, Foss A, Line PD, Scholz T, Jorgensen PF, Fosby B, Boberg KM, Mathisen O, Gladhaug IP, Egge TS, Solberg S, Hausken J, Dueland S. Liver transplantation for nonresectable liver metastases from colorectal cancer. Ann Surg. 2013 May;257(5):800-6. doi: 10.1097/SLA.0b013e3182823957. PMID 23360920
- [Background] Dueland S, Guren TK, Hagness M, Glimelius B, Line PD, Pfeiffer P, Foss A, Tveit KM. Chemotherapy or liver transplantation for nonresectable liver metastases from colorectal cancer? Ann Surg. 2015 May;261(5):956-60. doi: 10.1097/SLA.0000000000000786. PMID 24950280
- [Background] Gorgen A, Muaddi H, Zhang W, McGilvray I, Gallinger S, Sapisochin G. The New Era of Transplant Oncology: Liver Transplantation for Nonresectable Colorectal Cancer Liver Metastases. Can J Gastroenterol Hepatol. 2018 Jan 10;2018:9531925. doi: 10.1155/2018/9531925. eCollection 2018. PMID 29623268
- [Background] Fosby B, Melum E, Bjoro K, Bennet W, Rasmussen A, Andersen IM, Castedal M, Olausson M, Wibeck C, Gotlieb M, Gjertsen H, Toivonen L, Foss S, Makisalo H, Nordin A, Sanengen T, Bergquist A, Larsson ME, Soderdahl G, Nowak G, Boberg KM, Isoniemi H, Keiding S, Foss A, Line PD, Friman S, Schrumpf E, Ericzon BG, Hockerstedt K, Karlsen TH. Liver transplantation in the Nordic countries - An intention to treat and post-transplant analysis from The Nordic Liver Transplant Registry 1982-2013. Scand J Gastroenterol. 2015 Jun;50(6):797-808. doi: 10.3109/00365521.2015.1036359. PMID 25959101
- [Derived] Reivell V, Hagman H, Haux J, Jorns C, Lindner P, Taflin H. SOULMATE: the Swedish study of liver transplantation for isolated colorectal cancer liver metastases not suitable for operation or ablation, compared to best established treatment-a randomized controlled multicenter trial. Trials. 2022 Sep 30;23(1):831. doi: 10.1186/s13063-022-06778-9. PMID 36180944